CLINICAL TRIAL: NCT01591694
Title: National Child Traumatic Stress Network (NCTSN) Quality Improvement Initiative Database
Status: Completed | Type: Observational
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Principal Investigator, Harolyn M.E.Belcher, M.D., Director of Research, Kennedy Krieger Family Center; Associate Professor, Johns Hopkins University School of Medicine., Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Other Study IDs: NA_00047384; 2U79SM056215 (SAMHSA)
Record Dates: First submitted 2012-04-09; First posted 2012-05-04 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Post Traumatic Stress Disorder; Anxiety; Depression; Conduct Disorder; ADHD
Keywords: child trauma; maltreatment; physical abuse; sexual abuse; emotional abuse; abandonment; domestic violence; community violence
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression; Conduct Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- FamilyLive: Families with a history of intergenerational trauma (maltreatment, violence exposure, domestic violence, substance abuse, etc.)
- Yoga Based Psychotherapy: Children with a history of maltreatment and/or violence exposure
- Biofeedback: Children with a history of maltreatment and violence exposure and their caregivers
- TST-SA: Trauma Systems Therapy for Adolescent Substance Abuse

SUMMARY:
Trauma-informed treatment will improve emotional regulation and behavior.

DETAILED DESCRIPTION:
The proposed study is to request permission to continue federally mandated data collection to examine the clinical outcomes of children at the Family Center at Kennedy Krieger Institute who are enrolled in evidence-based and promising trauma-informed treatments as part of the National Child Traumatic Stress Network funded by the Substance Abuse and Mental Health Services Administration. The purpose of the National Child Traumatic Stress Initiative(NCTSNI) Evaluation is to determine the extent to which the NCTSI, through the National Child Traumatic Stress Network (NCTSN), has raised the standard of care and improved access to services for traumatized children. In addition, the evaluation assesses the extent to which the NCTSI has served as a national resource capable of improving children's access to high-quality, trauma-informed mental health services. This data, previously collected and managed by the Category I NCTSN Center at Duke will now be managed by ICF Macro in a data system entitled NICON.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled in treatment at the Family Center and caregivers

Exclusion Criteria:

* Psychosis,
* Inability to comply with directions

Ages: 2 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children enrolled in treatment at the Family Center and their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 4193 (Actual)
Dates: Start 2012-04; Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
Behavior | 1 year
  Improved behavioral and emotional regulation, i.e., improved behavior compliance, improved misbehavior symptoms, reduced symptoms of anxiety, depression, attention deficit hyperactivity disorder (ADHD), conduct disorder, oppositional defiant disorder, and post traumatic stress syndrome (PTSD). Improved sleep, toileting, parent-child attachment, and mood regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Harolyn Belcher, M.D., Principal Investigator — Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Locations (1):
- Family Center at Kennedy Krieger Institute, Baltimore, Maryland, United States